CLINICAL TRIAL: NCT00878345
Title: Dexmedetomidine Versus Pentobarbital Sedation Protocol for Non-painful Procedural Sedation in Pediatrics
Brief Title: Dexmedetomidine Versus Pentobarbital for Pediatric Procedural Sedation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never opened
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: colegroenersterni
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Sedation
Keywords: Pediatric sedation; Pentobarbital; Dexmedetomidine; Procedural sedation in children
MeSH Terms: interventions — Dexmedetomidine; Pentobarbital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Dexmedetomidine sedation protocol
  Interventions: Drug: dexmedetomidine sedation protocol
- 2 (Active Comparator): Pentobarbital sedation protocol
  Interventions: Drug: pentobarbital sedation protocol

INTERVENTIONS:
Drug: dexmedetomidine sedation protocol — Arm 1 will undergo sedation with dexmedetomidine, using 2 mcg/kg load IV over 10 minutes followed by an IV infusion of 1 mcg/kg/hr. May use versed 0.5 mg/kg IV x 1 for incomplete sedation, followed by increase of dexmedetomidine infusion to 1.5 mcg/kg/hr. Infusion will run throughout non-painful procedure (most likely MRI).
  Other Names: Precedex
  Arms: 1
Drug: pentobarbital sedation protocol — Pentobarbital Sedation Protocol IV: 2.5 mg/kg, followed by 1.25 mg/kg as needed x2. Maintenance: May give additional 1.25 mg/kg IV x 2 if needed. Max total dose of 200 mg pentobarbital throughout sedation.
  May give midazolam 0.05 mg/kg IV x 1 PRN agitation for rescue sedation.
  Other Names: Nembutal
  Arms: 2

SUMMARY:
The investigators believe dexmedetomidine will provide superior sedation with reduced side effects and reduced time to discharge compared with pentobarbital. The investigators have developed sedation protocols with pentobarbital and dexmedetomidine in our ambulatory procedure center. These protocols are both routinely used for sedation in our unit. The investigators propose to study these two protocols in children ages 6 months to 6 years presenting to the ambulatory procedure center for non-painful procedural sedation. The investigators will compare failure of sedation, side effect profile, recovery and discharge times between the two pharmacologic protocols.

ELIGIBILITY:
Inclusion Criteria:

* Requiring sedation for non-painful procedures
* Normal airway per exam

Exclusion Criteria:

* Congenital syndromes with known difficult airways
* Known difficult airway during past anesthesia or sedation experience
* Parent/guardian refusal of participation

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
failure of sedation | day of sedation

SECONDARY OUTCOMES:
side effect profile | 48 hours
post-sedation recovery and discharge time | day of sedation

CONTACTS AND LOCATIONS:
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Mason KP, Zgleszewski SE, Prescilla R, Fontaine PJ, Zurakowski D. Hemodynamic effects of dexmedetomidine sedation for CT imaging studies. Paediatr Anaesth. 2008 May;18(5):393-402. doi: 10.1111/j.1460-9592.2008.02451.x. Epub 2008 Mar 18. PMID 18363628
- [Background] Mukhtar AM, Obayah EM, Hassona AM. Preliminary experience with dexmedetomidine in pediatric anesthesia. Anesth Analg. 2006 Jul;103(1):250. doi: 10.1213/01.ANE.0000228303.92422.73. No abstract available. PMID 16790665
- [Background] Koroglu A, Teksan H, Sagir O, Yucel A, Toprak HI, Ersoy OM. A comparison of the sedative, hemodynamic, and respiratory effects of dexmedetomidine and propofol in children undergoing magnetic resonance imaging. Anesth Analg. 2006 Jul;103(1):63-7, table of contents. doi: 10.1213/01.ANE.0000219592.82598.AA. PMID 16790627